CLINICAL TRIAL: NCT04278859
Title: A Phase I Clinical Study of JS004, a Recombinant Humanized mAb Specific to B-and T-Lymphocyte Attenuator (BTLA), in Subjects With Advanced Solid Malignancies
Brief Title: Safety, Tolerability and Pharmacokinetics of a Recombinant Humanized mAb Specific to B-and T-Lymphocyte Attenuator (BTLA) for Injection in Subjects With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JS004-001-I
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0.3mg/kg repeat dose every 21 days up to 2 years (Experimental)
  Interventions: Biological: Drug: JS004, Recombinant humanized IgG4κ monoclonal antibody specific to BTLA for injection Intravenous infusion
- 1 mg/kg repeat dose every 21 days up to 2 years; (Experimental)
  Interventions: Biological: Drug: JS004, Recombinant humanized IgG4κ monoclonal antibody specific to BTLA for injection Intravenous infusion
- 3 mg/kg repeat dose every 21 days up to 2 years; (Experimental)
  Interventions: Biological: Drug: JS004, Recombinant humanized IgG4κ monoclonal antibody specific to BTLA for injection Intravenous infusion
- 10 mg/kg repeat dose every 21 days up to 2 years; (Experimental)
  Interventions: Biological: Drug: JS004, Recombinant humanized IgG4κ monoclonal antibody specific to BTLA for injection Intravenous infusion

INTERVENTIONS:
Biological: Drug: JS004, Recombinant humanized IgG4κ monoclonal antibody specific to BTLA for injection Intravenous infusion — Drug: JS004, Recombinant humanized IgG4κ monoclonal antibody specific to BTLA for injection Intravenous infusion
  Other Names: TAB004

SUMMARY:
A 3-part (dose-escalation, dose-expansion and cohort-expansion) phase I clinical study of JS004 in subjects with advanced solid malignancies in China for the first time, to evaluate the safety, tolerability, PK, immunogenicity, antitumor activity and biomarkers of JS004, define the MTD and RP2D. A cycle is 21 days (3 weeks) which includes JS004 being administered IV Q3W. All patients will be treated until disease progression per RECIST v1.1 and iRECIST, or intolerable toxicity per CTCAE 5.0, withdrawal of consent, or end of the study, whichever occurs first.Disease progression must be confirmed at least 4 weeks but no longer than 8 weeks after initial documentation of progression.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and willing to sign the Informed Consent Form;
2. 18-70 years(included), male or female;
3. Subjects with histologically or cytologically confirmed advanced solid tumor.
4. In Dose Escalation and Dose Expansion, patients must have received, or be ineligible for or intolerant of all available approved or standard therapies known to confer clinical benefit, or for whom no standard therapy exists; in Indication Extension, patients with advanced solid tumors, who must have received at least one line of therapy for advanced or metastatic disease, but are not required to have received all standard therapies known to confer clinical benefit;
5. ECOG performance status of 0 or 1;
6. Life expectancy ≥12 weeks;
7. At least one measurable lesion per RECISTv1.1 and iRECIST;
8. Willingness to provide consent for fresh pre-treatment biopsies, or,an archival specimen could be required within two years prior to the first dose of study drug;
9. Adequate organ and marrow function per protocol specifically defined;
10. Females of childbearing potential ,and males who are sexually active with a female partner of childbearing potential, must use effective contraception from time of screening, and must agree to continue using such precautions for 3 months after the final dose of JS004; HCG testing will be conducted and negative result within 7 days before randomization for females of childbearing potential, and must not be breast-feeding;

Exclusion Criteria:

1. Known allergic reaction to any monoclonal antibody or the ingredients and compositions of JS004 .
2. Prior exposure to anti-BTLA, or anti-HVEM antibodies.
3. Concurrent enrollment in another clinical study within 4 weeks prior to first dose of JS004, unless it is an observational (non-interventional) clinical study or the follow-up period of an interventional study.
4. Major surgery (as defined by the investigator) within 4 weeks prior to first dose of JS004 or still recovering from prior surgery.Any concurrent chemotherapy within 4 weeks prior to first dose of JS004 , radiotherapy, immunotherapy, or biologic therapy for cancer treatment. Traditional Chinese/Chinese Patent Medicine preparations within 2 weeks prior to first dose of JS004 for treating tumors approved by NMPA.Concurrent use of hormones for non-cancer-related conditions (e.g., insulin for diabetes and hormone replacement therapy) is acceptable. Isolated lesions for palliative intent is acceptable (e.g., by local surgery or radiotherapy) without influence in efficacy assessment.
5. Patients who have discontinued prior immune therapy due to immune mediated adverse reaction(s).
6. Current or prior use of immunosuppressive medication within 4 weeks prior to the first dose of JS004, with the exception of intranasal and inhaled corticosteroids or systemic corticosteroids not to exceed 10 mg/day of prednisone or equivalent.
7. Prior allogeneic bone marrow transplantation or prior solid organ transplantation.
8. Receipt of live attenuated vaccination within 30 days of receiving JS004.
9. Two or more malignant tumors within 5 years prior to the first dose of JS004. Except the following conditions: radically cured early malignant tumor (carcinoma in situ or stage I tumor), for example, adequately treated cervical carcinoma in situ, basal or squamous cell skin cancer.
10. Symptomatic or untreated central nervous system (CNS) metastases or requiring ongoing treatment for CNS metastases, including corticosteroids and antiepileptic agents. Subjects with previously treated brain metastases may participate unless clinically stable for at least 4 weeks prior to study entry, have no evidence of new or enlarging metastases, and are off steroids.
11. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to baseline or to NCI-CTCAE v5.0 Grade 0 or 1, or to levels dictated in the inclusion/exclusion criteria with the exception of alopecia. Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by JS004 may be included (e.g., hearing loss) after consultation with the medical monitor.
12. Active or prior documented autoimmune disease, such as but not limited to systemic lupus erythematosus or multiple sclerosis, within the past 2 years.
13. History of anaphylaxis, eczema that cannot be controlled with topical corticosteroids, or asthma.
14. History of primary immunodeficiency.
15. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, fever of unknown origin > 38.5 °C ( Subjects with tumorous fever will be determined by investigator), symptomatic congestive heart failure according to New York Heart Association (NYHA) Functional Classification ≥ 3, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis
16. Patients with known history of active tuberculosis, and drug-induced interstitial lung disease or pneumonitis ≥ Grade 2.
17. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
18. Subjects who are known to be human immunodeficiency virus (HIV) positive.
19. Subjects with evidence of hepatitis B or C virus infection, unless their hepatitis is considered to have been cured. (Note that subjects with prior hepatitis B virus [HBV] infection, HBc Ab positive and HBs Ag negative at screening visit, must have HBV viral load [VL] less than the local normal range of study site before study enrollment; hepatitis C virus [HCV] infection must have, HCV RAV negative before study enrollment.
20. Pregnant or breastfeeding women.
21. Patients with vitiligo, alopecia and controlled endocrine deficiency by hormone replacement therapy, such as hypothyroidism, can be included. Patients with rheumatoid arthritis and other joint diseases, Schering's syndrome, chylosis and psoriasis that have been controlled with topical administration, and patients with positive serological tests such as antinuclear antibody (ANA) and antithyroid antibody, should be assessed whether target organs are affected and systemic treatment required. It is up to the investigator to determine if the patient could be enrolled or not.
22. Having other factors that may possibly cause halfway-termination of this study as judged by investigators, for example, which may influence the right & benift、safety of subjects, incompliance with the protocol, the capability to be informed consent, and other medical (e.g. the conditions or disease of respiratory, metabolic, congenital, endocrine and central nervous system, etc), family or social factors.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2023-07-13 (Actual)

PRIMARY OUTCOMES:
DLT, MTD, Number of participants and severiaty with treatment-related Adverse events (AEs) as assessed by CTCAE v5.0 | 2 years
  DLT, MTD, Number of participants and severity with treatment-related Adverse events (AEs) as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
ORR | 2 years
  Objective Response Rate(ORR) by RECIST 1.1
DOR | 2 years
  Duration of Response (DOR) by RECIST 1.1
DCR | 2 years
  Disease Control Rate (DCR) by RECIST 1.1
PFS | 2 years
  Progression-free survival(PFS) by RECIST 1.1
OS | 2 years
  Overall survival(OS) by RECIST 1.1
RO | 2 years
  BTLA receptor of occupancy (RO) of blood
Cmax | 2 years
  Maximum Plasma Concentration(Cmax) after injection of JS004
Tmax | 2 years
  Perk Time(Tmax) after injection of JS004
Area Under the Cure(AUC) after injection of JS004 | 2 years
  AUC
t1/2 half life | 2 years
  t1/2 after injection of JS004
Plasma Clearance(CL) | 2 years
  Plasma Clearance(CL) after injection of JS004
Volume of distribution(V) | 2 years
  Apparent volume of distribution after injection of JS004
Cmin | 2 years
  Minimum Plasma concentration(Cmin) of steady state after multiple dose injection of JS004
volume of distribution of steady state (Vss) | 2 years
  Apparent volume of distribution of steady state (Vss) after multiple dose injection of JS004
ADA | 2 years
  The presence of anti-drug antibody (ADA) after multiple dose injection of JS004

OTHER OUTCOMES:
Predictive biomarkers | 2 years
  Predictive biomarkers, including but not limited to, BTLA and HVEM

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijin, Beijing Municipality, China